CLINICAL TRIAL: NCT02756130
Title: A Phase I/II, Single Center, Proof-of-Concept Study of Birinapant in Combination With Platinum Based Chemotherapy Targeting Recurrent High Grade Serous Ovarian Carcinomas (HGSOC)
Brief Title: Birinapant and Carboplatin in Treating Patients and Targeting Recurrent High Grade Ovarian, Fallopian Tube, or Primary Peritoneal Cancer (HGSOC)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: funding was not secured
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other); TetraLogic Pharmaceuticals (Industry); Alpha Stem Cell Clinic (ASCC) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-000746; NCI-2016-00596 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GODL001 (Other: Jonsson Comprehensive Cancer Center); 16-000746 (Other: UCLA / Jonsson Comprehensive Cancer Center); NCT03027271 (obsolete NCT alias)
Record Dates: First submitted 2016-04-22; First posted 2016-04-29 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2018-08

CONDITIONS: High Grade Fallopian Tube Serous Adenocarcinoma; High Grade Ovarian Serous Adenocarcinoma; Primary Peritoneal High Grade Serous Adenocarcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — birinapant; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (birinapant, carboplatin) (Experimental): Patients receive birinapant IV over 30 minutes on days 1 and 8, and carboplatin IV over 30 minutes to 1 hour on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Birinapant; Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Birinapant — Given IV
  Other Names: TL32711
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I/II trial studies how well birinapant and carboplatin work in treating patients with ovarian, fallopian tube, or primary peritoneal cancer that has come back. Drugs used in chemotherapy, such as birinapant and carboplatin work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether addition of birinapant to carboplatin therapy can reduce the percentage of platinum resistant tumor initiating cells by 50% compared to pre-therapy biopsies in participants with recurrent high grade serous ovarian carcinomas (HGSOC) whose tumors score positive in the in vitro organoid bioassay test.

II. Assess target engagement by comparing levels of cellular inhibitor of apoptosis protein (cIAP) and percentage of apoptotic cells in pre-versus post therapy tumor biopsies (obtained after three cycles of treatment).

SECONDARY OBJECTIVES:

I. To see if there is an increase in progression free survival of participants treated with co-therapy (birinapant/carboplatin) compared with historic controls.

TERTIARY OBJECTIVES:

I. Develop a companion diagnostic test by correlating clinical response seen in participants with two biomarker assays developed in our laboratory.

1. Measuring levels of cIAP protein by western blot in tumor biopsies obtained from participants prior to start of therapy.
2. Measuring percentage of cIAP positive cells by immunohistochemistry in tumor biopsies obtained from participants prior to start of therapy.

OUTLINE:

Patients receive birinapant intravenously (IV) over 30 minutes on days 1 and 8, and carboplatin IV over 30 minutes to 1 hour on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 2 years from Course 1, Day 1.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have measurable disease by imaging defined as tumor that can be measured >= 10 mm with multiparametric magnetic resonance imaging (MRI) (primary modality of imaging) or computed tomography (CT) (as an alternative) or >= 10 mm by caliper on physical examination
* Participant is capable of understanding and complying with parameters as outlined in the protocol and able to sign and date the informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to initiation of any screening or study-specific procedures
* The participant must have a histologic diagnosis of recurrent high grade serous ovarian cancer (ovarian, tubal, peritoneal), to be treated with chemotherapy
* Participants must have an image guided biopsy performed to yield fresh tissue for the in vitro organoid bio-assay and two biomarker testing (western blot and immunohistochemistry)
* Only patients with tumors that score positive in the in vitro organoid bio-assay will be enrolled in the clinical trial; patients with tumors that score negative in this bio-assay will be considered screening failures and will not be enrolled in the clinical trial
* Participant must have either no neuropathy (sensory and motor) or neuropathy less than or equal to grade 1
* The participant must have an Eastern Cooperative Oncology Group (ECOG) score between 0 - 2 at screening
* The participant must have a life expectancy of greater than 12 weeks
* Absolute neutrophil count >= 1,500/mm^3
* Platelets >= 100,000/ mm^3
* Hemoglobin >= 9 g/dL or equivalent
* Total bilirubin =< 1.5 ? institutional upper limit of normal (ULN), unless known Gilbert?s syndrome has been diagnosed
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 ? institutional ULN (=< 5 ? ULN if liver metastasis)
* Serum creatinine =< 1.5 ? ULN or creatinine clearance >= 50 mL/min/1.73 m^2
* Amylase < ULN
* Lipase < ULN
* Female participants of childbearing potential must have a negative serum pregnancy test at screening and negative (serum or urine) pregnancy test within 72 hours before the first study-drug dose; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required; the serum pregnancy test must be negative for the participant to be eligible
* Female participants of childbearing potential should ensure use of a highly effective method of birth control as defined by the investigator, for example, those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectable, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomized partner during the study and for a period of at least 4 months following the last dose of any drug administered during the study

Exclusion Criteria:

* Patients with tumors that score negative in the in vitro organoid bio-assay will be excluded
* Patients with non-measurable disease < 10 mm on multiparametric MRI or CT scan will be excluded
* Participants with a secondary malignancy that is progressing or requires active treatment; participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or in situ cervical cancer that has undergone potentially curative treatment are not excluded
* Participants who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to birinapant or its constituents
* Participants requiring the use of anti-tumor necrosis factor (anti-TNF) therapies, such as infliximab, or has received treatment with anti-TNF therapies within 5 half-lives of the drug
* Participants with an uncontrolled inter-current illness including, but not limited to, symptomatic congestive heart failure, hypertension, unstable angina pectoris, cardiac arrhythmia, autoimmune disease or inflammatory diseases, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women or women who expect to conceive a child are excluded from the study; breastfeeding should be discontinued if the mother is treated on this study
* Participants who have a known active infection requiring systemic therapy, including human immunodeficiency virus (HIV), hepatitis B, and hepatitis C
* Participants with a history of cranial nerve palsy
* Participant is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is an investigational site or sponsor-investigator staff directly involved with this trial, unless prospective IRB approval (by chair or designee) is granted allowing exception to this criterion for a specific subject
* In the opinion of the investigator, the participant is an unsuitable candidate for this study
* Patients who are taking or anticipate taking any maintenance therapy while actively being treated on protocol or while being followed on protocol will be excluded; an example of this would be maintenance therapy with a Poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibitor such as olaparib

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in percentage of cancer initiating cells | Baseline up to 2 years
  Will be measured using a 3-dimensional organoid assay; population analysis using flow cytometry to measure the overall percentage of platinum resistant tumor initiating cells and by immunohistochemistry. Percent cellular inhibitor of apoptosis (cIAP) positive and amount of cIAP protein will be computed using either the non parametric Wilcoxon signed rank test or the paired t test if the data follow a normal distribution. Full summary statistics including the mean and median difference and the corresponding 95% confidence bounds will be reported. We will report scatter plots and the non parametric Spearman correlation coefficients among these four measures of platinum resistant tumor initiating cells pre-therapy as well as the post- minus pre-treatment difference.
Pharmacodynamic analysis of cellular inhibitor of apoptosis (cIAP) protein | Baseline up to 2 years
  Will measure the level of cIAP protein in pre- versus (vs). post-therapy tumors, measured by quantitative western blot, compared to a purified cIAP standard of known amount loaded on the same gel. Percent cIAP positive and amount of cIAP protein will be computed using either the non parametric Wilcoxon signed rank test or the paired t test if the data follow a normal distribution. Full summary statistics including the mean and median difference and the corresponding 95% confidence bounds will be reported. We will report scatter plots and the non parametric Spearman correlation coefficients among these four measures of platinum resistant tumor initiating cells pre-therapy as well as the post- minus pre-treatment difference.

SECONDARY OUTCOMES:
Progression free survival (PFS) assessed using imaging (multiparametric magnetic resonance imaging [MRI] (primary modality of imaging) of computed tomography (CT) and the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria | Start of therapy and progression of disease or death whichever comes first, assessed up to 2 years
  The secondary analysis in each group will be comparison of PFS to known historical PFS. The PFS curve will be estimated using the Kaplan-Meier method and the sample PFS curve will be compared to the known historical population curve using the one sample log rank test.

OTHER OUTCOMES:
Cellular inhibitor of apoptosis (cIAP) expression by immunohistochemistry with patient response to co-therapy | Up to 2 years
  Evaluated using non parametric receiver operator characteristic (ROC) methods with the corresponding accuracy statistics reported.
Cellular inhibitor of apoptosis (cIAP) expression by western blot with patient response to co-therapy | Up to 2 years
  Evaluated using non parametric ROC methods with the corresponding accuracy statistics reported.

CONTACTS AND LOCATIONS:
Overall Officials: Sanaz Memarzadeh, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States